CLINICAL TRIAL: NCT03195790
Title: Value and Mechanisms of Home Visitation in Obesity Interventions for Low-income Children
Brief Title: Creating Healthy Environments for Chicago Kids
Acronym: CHECK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15120306; R01DK111358 (NIH)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessors, PI, and some co-investigators will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical center treatment arm (Active Comparator): Family-based pediatric obesity treatment delivered at an urban medical center.
  Interventions: Behavioral: Family-based pediatric obesity treatment
- Home treatment arm (Experimental): Family-based pediatric obesity treatment delivered in the family's home.
  Interventions: Behavioral: Family-based pediatric obesity treatment

INTERVENTIONS:
Behavioral: Family-based pediatric obesity treatment — Families with at least one overweight/obese child between ages 6 and 11 years will receive 12-months of family-based pediatric obesity treatment that emphasizes healthy changes to the home environment and family routines. The intervention targets dietary intake, physical activity, and consistent sleep.

SUMMARY:
Pediatric obesity interventions for low-income populations are increasingly delivered in children's homes, which may make treatment more accessible to families and enhance the potency of the intervention in several ways. This randomized trial will directly test whether delivering family-based behavioral interventions for pediatric overweight/obesity in the home setting improves weight loss outcomes in low-income children relative to medical center-based treatment. The trial will also quantify the cost-effectiveness of home visitation, and explore the mechanisms accounting for observed treatment effects

DETAILED DESCRIPTION:
The goal of this project is to systematically evaluate the incremental weight loss benefit and cost-effectiveness of delivering standard family-based treatment for pediatric overweight/obesity in the home setting vs. traditional medical settings. In a randomized controlled trial involving low-income households, 266 children ages 6-12 years will be allocated to 12 months of family-based treatment delivered either in their home or at an urban academic medical center. Both arms will receive the same intervention content and dosage, and differ only in the location of in-person treatment sessions. Aim 1 is to test the hypothesis that home-based treatment produces a greater reduction in child adiposity, reflected in 12-month change in BMI z-score. Aim 2 is to compare the cost-effectiveness of home-based treatment to medical center-based treatment, and calculate the added cost of the incremental weight loss benefit associated with home visitation. These data will inform efforts to disseminate home-based interventions for low-income populations by public health agencies and third-party payers. Aim 3 is to explore specific mechanisms through which home visitation may improve weight loss outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Family includes at least one child who is 6 to 12 years old, and is overweight or obese (has a body mass index at or above the 85th percentile for age and sex)
* Child's household has an income-to-poverty ratio ≤ 2.0

Exclusion Criteria:

* Child or caregiver(s) are not fluent in English
* Unwilling to attend and complete either home-based or clinic-based treatment, or to complete any aspect of the study assessment battery
* Medical contraindication or barrier to weight loss treatment
* Caregiver has a major medical or psychiatric condition likely to interfere with treatment
* Plans to relocate outside the Chicago area in the next 12 months, or living in temporary or group housing with other families
* Resides more than 15 miles from the Illinois Medical District (study site)
* Conditions in or around the home that jeopardize staff/interventionist safety

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Child adiposity | 12 months
  Change from baseline in child body mass index z-score (zBMI)

SECONDARY OUTCOMES:
Clinically significant weight loss | 12 months
  Proportion of children achieving adiposity reduction of at least 0.25 zBMI
Cost-effectiveness | 12 months
  Incremental cost-effectiveness ratio of home-based vs medical center treatment, calculated from societal perspective.

OTHER OUTCOMES:
Intervention dosage | 12 months
  Dosage of intervention received in each arm, in units of clock time of intervention delivered
Treatment recommendations | 12 months
  Number of specific treatment recommendations provided to each family
Change in the home food environment | 12 months
  Number of obesity-promoting foods and beverages present in the home, measured by staff audits
Change in the home physical activity and media environment | 12 months
  Sports equipment and media devices in the home, measured by staff audits
Change in family routines | 12 months
  Family routines associated with childhood obesity risk, assessed through the Family Nutrition and Physical Activity Screening Tool

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
This plan is to be determined.

REFERENCES:
- [Derived] Appelhans BM, French SA, Bradley LE, Lui K, Janssen I, Richardson D. CHECK: A randomized trial evaluating the efficacy and cost-effectiveness of home visitation in pediatric weight loss treatment. Contemp Clin Trials. 2020 Jan;88:105891. doi: 10.1016/j.cct.2019.105891. Epub 2019 Nov 15. PMID 31740429

DOCUMENTS (1):
  • Informed Consent Form (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03195790/ICF_000.pdf